CLINICAL TRIAL: NCT00767949
Title: A Phase 1, Dose-Escalating, Multi-Center, Study of iSONEP (Sonepcizumab [LT1009]) Administered as an Intravitreal Injection to Subjects With Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Safety Study of iSONEP (Sonepcizumab/LT1009) to Treat Neovascular Age-related Macular Degeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lpath, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT1009-Oph-001
Record Dates: First submitted 2008-10-02; First posted 2008-10-07 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: wet; AMD
MeSH Terms: interventions — sonepcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): iSONEP
  Interventions: Biological: iSONEP

INTERVENTIONS:
Biological: iSONEP — single intravitreal injection of 0.2, 0.6, 1.0, 1.4 or 1.8 mg/eye
  Other Names: Sonepcizumab; LT1009

SUMMARY:
Age-related macular degeneration (AMD) is a disease that, in time, destroys the macula, which is the central part of the retina that gives sharp central vision. The primary purpose of this study is to assess the safety of iSONEP which is a humanized monoclonal antibody against a bioactive lipid, sphingosine 1-phosphate (S1P).

DETAILED DESCRIPTION:
S1P modulates the AMD-associated processes of angiogenesis, inflammation and fibrosis. A potential strategy for treating choroidal neovascularization associated with AMD is to reduce the biologically available extracellular levels of S1P. iSONEP is highly selective for S1P and binds with picomolar affinity. Lpath proposes that iSONEP would deprive many cell types (fibroblasts, pericytes, vascular endothelial cells and inflammatory) of important growth and survival factors thus targeting the multiple maladaptive processes of exudative AMD that ultimately result in the loss of photoreceptors, their supporting cells, and visual acuity. Targeting simultaneously multiple components of the choroidal neovascular response is a novel approach and has the potential to be more potent than "single-targeted" therapeutics such as anti-VEGF therapies.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older
* BCVA ETDRS letter score in study eye between 20-57 letters using ETDRS refraction (Snellen of 20/70-20/400)
* Any CNV secondary to AMD in study eye, classic, minimally classic or occult with leakage on fluorescein angiography and intraretinal or subretinal fluid on OCT
* Visual acuity in fellow eye must be 20/800 or better at 4 meters
* Able to read, understand and sign the consent form before entering into study

Exclusion Criteria:

* Ocular disease other than CNV that could compromise vision in study eye
* Systemic immunosuppressive medication/therapy (e.g., chemotherapy, steroids)
* Uncontrolled hypertension and/or arrhythmias
* QT/QTc interval measurement >450 msec
* Cancer within the last 2 years except superficial basal or squamous cell skin cancer or cervical carcinoma in situ
* Have angioid streaks, presumed ocular histoplasmosis syndrome, myopia (>8 diopters) or CNV secondary to other causes than AMD
* Any additional ocular diseases which have irreversibly compromised visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema and severe non-proliferative diabetic retinopathy
* Any intraocular or general surgery, including cataract surgery, within 2 months of Day 1
* History of uveitis in either eye
* Any ocular or periocular infection within 4 weeks prior to Day 1
* Active ocular inflammation grade trace and above
* Cup to disc ratio >0.8, IOP >21 mmHg in glaucoma subjects treated with more than 2 ocular hypotensive agents
* Previous pars plana vitrectomy or trabeculectomy in study eye
* History of anterior vitrectomy
* Inability to obtain photographs, FA or OCT to document CNV, e.g. due to media opacity, allergy to fluorescein dye or lack of venous access
* Aphakia
* Previous intravitreal Macugen, Avastin or Lucentis (injection or drug device implantation) in study eye within 6 weeks or triamcinolone within 6 months
* Receiving or requiring chronic concomitant therapy with systemic anti-angiogenic treatments p.o., parenteral (excluding inhaled steroids) (>5 mg) or topical corticosteroids in the study eye
* PDT within 12 weeks prior to Day 1
* Subjects taking systemic anticoagulants such as warfarin
* Investigational agents or devices within 6 weeks prior to Day 1
* Females who are pregnant or nursing and women of child bearing potential who are not using adequate contraceptive precautions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To determine safety, tolerability, maximum tolerated dose and dose-limiting toxicity of iSONEP following a single intravitreal injection to subjects with choroidal neovascularization secondary to AMD | Active phase: 30 days post-injection; Follow-up phase: 12 months post-injection

SECONDARY OUTCOMES:
To characterize systemic pharmacokinetics, evaluate the immunogenicity, and investigate preliminary efficacy on retinal lesion thickness determined by OCT; size and extent of CNV and lesion area; and visual acuity | Active phase: 30 days post-injection; Follow-up phase: 12 months post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Stoller, MD, Study Director — Lpath, Inc.
Locations (5):
- United States (5):
  - Retinal Consultants of Arizona, LTD, Phoenix, Arizona
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Vitreo-Retinal Consultants, Grand Rapids, Michigan
  - Wills Eye Institute, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Visentin B, Vekich JA, Sibbald BJ, Cavalli AL, Moreno KM, Matteo RG, Garland WA, Lu Y, Yu S, Hall HS, Kundra V, Mills GB, Sabbadini RA. Validation of an anti-sphingosine-1-phosphate antibody as a potential therapeutic in reducing growth, invasion, and angiogenesis in multiple tumor lineages. Cancer Cell. 2006 Mar;9(3):225-38. doi: 10.1016/j.ccr.2006.02.023. PMID 16530706
- [Background] Caballero S, Swaney J, Moreno K, Afzal A, Kielczewski J, Stoller G, Cavalli A, Garland W, Hansen G, Sabbadini R, Grant MB. Anti-sphingosine-1-phosphate monoclonal antibodies inhibit angiogenesis and sub-retinal fibrosis in a murine model of laser-induced choroidal neovascularization. Exp Eye Res. 2009 Mar;88(3):367-77. doi: 10.1016/j.exer.2008.07.012. Epub 2008 Aug 6. PMID 18723015